CLINICAL TRIAL: NCT03410524
Title: Simethicone Pretreatment With Low-volume Polyethylene Glycol-3350 and Bisacodyl in an Effort to Improve Bowel Wall Visualization During Colonoscopy
Brief Title: Evaluation of Oral Simethicone With Low Volume Polyethylene Glycol Bowel Preparation During Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Collaborators: Gastroenterology Consultants (Unknown)
Responsible Party: Principal Investigator, Mohit Rishi, Resident physician - Department of Internal Medicine, University of Nevada, Reno
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1139179
Record Dates: First submitted 2018-01-09; First posted 2018-01-25 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Colonoscopy
Keywords: Bowel wall visualization; Intraluminal bubbles; Intraluminal foam; Simethicone
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Endoscopist and patient blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simethicone with PEG-3350 bisacodyl preparation (Active Comparator): Treatment arm:
  200 mg Simethicone in 3 mL of liquid formulation mixed with low volume PEG-3350 bisacodyl combination preparation. Bowel preparation taken as per directions including the evening before and the day of the procedure.
  Interventions: Drug: Simethicone Solution
- Placebo with PEG-3350 bisacodyl preparation (Placebo Comparator): Placebo arm:
  3 mL of water mixed with low volume PEG-3350 bisacodyl combination preparation. Bowel preparation taken as per directions including the evening before and the day of the procedure.
  Interventions: Drug: Water

INTERVENTIONS:
Drug: Simethicone Solution — 200 mg of Simethicone in 3 mL of Simethicone Solution Formulation
  Arms: Simethicone with PEG-3350 bisacodyl preparation
Drug: Water — 3 mL of water as placebo added to the bowel preparation
  Arms: Placebo with PEG-3350 bisacodyl preparation

SUMMARY:
An adequate bowel preparation has been well established to lead to a successful colonoscopy. Research has consistently demonstrated inadequate bowel preparation with lower adenoma detection rates. Over the years, endoscopy centers have changed the constituents of bowel preparation in light of new research. In 2006, 3 medical organizations recommended the use of polyethylene glycol (PEG) solution for bowel preparation. Initially, a 4 liter PEG solution was commonly used using a split dose regimen for bowel prep. However, many patients found that this large volume gave them side effects including bloating and cramping. Other studies showed that a low volume PEG solution with oral bisacodyl fared equally in terms of adequacy of bowel preparation. With the institution of lower volume PEG preparation our offices noted improved patient toleration, satisfaction, and clinical outcomes. However, multiple endoscopists have noticed an increased in intraluminal bubbles and foam with the low volume preparation. This can impair proper visualization of the bowel wall even with an adequate bowel preparation. The current standard of practice includes irrigation, lavage, and suctioning using a simethicone infused saline during the colonoscopy. Its property of reducing surface tension to help dissolve bubbles and clear the field of view is vital during the procedure. Furthermore, it does not dissolve into the blood stream and thereby, is considered rather safe.

This study evaluates whether the addition of oral simethicone with the colonoscopy bowel preparation reduces bubbles and foam during the procedure using a randomized and controlled interventional study.

DETAILED DESCRIPTION:
This prospective, multi-center, randomized, controlled, double (patient and endoscopist) blinded study is conducted at the Gastroenterology Consultants outpatient clinics and endoscopy centers in association with the University of Nevada-Reno School of Medicine. After obtaining signed informed consent, outpatients are recruited and randomized into 1 of 2 treatment groups; PEG3350-Bisacodyl with 200 mg liquid simethicone treatment and PEG3350-Bisacodyl treatment with inert placebo (water).

The primary outcome includes reduction of bubbles using the intraluminal bubbles scale. Secondary outcomes include the evaluations of the numbers and types of polyps, numbers and types of masses detected, cecal insertion time, withdrawal time, adverse effects, and the adequacy of bowel prep using the Boston Bowel Prep scale.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for outpatient elective colonoscopy
* Adult 18-80 years of age able to give consent.
* English speaking adults.

Exclusion Criteria:

* History of bowel resection
* Uncontrolled hypertension
* Suspected bowel perforation
* Suspected bowel obstruction
* Indications for emergent/urgent colonoscopy
* Non-english speaking individuals

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Intraluminal Bubbles Scale | Data reported during colonoscopy.
  I >90% of the mucosal circumference seen II 90%-75% of the mucosal seen without foam or bubbles not requiring irrigation III 74% to 50% of the mucosa is free of foam or bubbles. Required irrigation IV <50% of the mucosa seen free of foam or bubbles. Required irrigation

SECONDARY OUTCOMES:
Boston Bowel Preparation Scale | Data reported during colonoscopy.
Cecal insertion time | Data reported during colonoscopy.
Withdrawal time | Data reported during colonoscopy.
Number of polyp | Data reported during colonoscopy.
Type of polyp | Post colonoscopy pathology. Up until pathology data reporting. Estimated up to 2 weeks after colonoscopy.
Type of masses | Post colonoscopy pathology. Up until pathology data reporting. Estimated up to 2 weeks after colonoscopy.
Number of masses | Data reported during colonoscopy.
Adverse effects | From the time of administration of the bowel preparation (day prior to colonoscopy) up until the time of the procedure preparation (pre-colonoscopy preparation). Estimated period of up to 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Osgard, MD, Principal Investigator — University of Nevada School of Medicine
Locations (2):
- United States (2):
  - Gastroenterology Consultants Reno - North Office and Endoscopy Center, Reno, Nevada
  - Gastroenterology Consultants Reno - South Meadows Office and Endoscopy Center, Reno, Nevada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kojecky V, Matous J, Keil R, Dastych M, Kroupa R, Zadorova Z, Varga M, Dolina J, Kment M, Hep A. A head-to-head comparison of 4-L polyethylene glycol and low-volume solutions before colonoscopy: which is the best? A multicentre, randomized trial. Int J Colorectal Dis. 2017 Dec;32(12):1763-1766. doi: 10.1007/s00384-017-2901-x. Epub 2017 Sep 24. PMID 28944412
- [Background] Parmar R, Martel M, Rostom A, Barkun AN. Validated Scales for Colon Cleansing: A Systematic Review. Am J Gastroenterol. 2016 Feb;111(2):197-204; quiz 205. doi: 10.1038/ajg.2015.417. Epub 2016 Jan 19. PMID 26782820
- [Background] Parente F, Vailati C, Bargiggia S, Manes G, Fontana P, Masci E, Arena M, Spinzi G, Baccarin A, Mazzoleni G, Testoni PA. 2-Litre polyethylene glycol-citrate-simethicone plus bisacodyl versus 4-litre polyethylene glycol as preparation for colonoscopy in chronic constipation. Dig Liver Dis. 2015 Oct;47(10):857-63. doi: 10.1016/j.dld.2015.06.008. Epub 2015 Jul 6. PMID 26232311
- [Background] Tongprasert S, Sobhonslidsuk A, Rattanasiri S. Improving quality of colonoscopy by adding simethicone to sodium phosphate bowel preparation. World J Gastroenterol. 2009 Jun 28;15(24):3032-7. doi: 10.3748/wjg.15.3032. PMID 19554657
- [Background] American Society of Colon and Rectal Surgeons (ASCRS); American Society for Gastrointestinal Endoscopy (ASGE); Society of American Gastrointestinal and Endoscopic Surgeons (SAGES); Wexner SD, Beck DE, Baron TH, Fanelli RD, Hyman N, Shen B, Wasco KE. A consensus document on bowel preparation before colonoscopy: prepared by a Task Force from the American Society of Colon and Rectal Surgeons (ASCRS), the American Society for Gastrointestinal Endoscopy (ASGE), and the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES). Surg Endosc. 2006 Jul;20(7):1161. doi: 10.1007/s00464-006-3037-1. No abstract available. PMID 16799744
- [Background] Adams WJ, Meagher AP, Lubowski DZ, King DW. Bisacodyl reduces the volume of polyethylene glycol solution required for bowel preparation. Dis Colon Rectum. 1994 Mar;37(3):229-33; discussion 233-4. doi: 10.1007/BF02048160. PMID 8137669
- [Background] Harrison NM, Hjelkrem MC. Bowel cleansing before colonoscopy: Balancing efficacy, safety, cost and patient tolerance. World J Gastrointest Endosc. 2016 Jan 10;8(1):4-12. doi: 10.4253/wjge.v8.i1.4. PMID 26788258
- [Background] Brecevic L, Bosan-Kilibarda I, Strajnar F. Mechanism of antifoaming action of simethicone. J Appl Toxicol. 1994 May-Jun;14(3):207-11. doi: 10.1002/jat.2550140311. PMID 8083482